CLINICAL TRIAL: NCT01180491
Title: A Clinical Investigation on Early Visible Effects of Application of K101 During 8 Weeks on Discoloured and Deformed Nails Resulting From Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moberg Pharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: K101-50
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Onychomycosis
Keywords: Discoloured and deformed nails resulting from onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: K101 nail solution

SUMMARY:
The purpose of this study is to further evaluate and document early visible effects on nail appearance of topical K101.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older
* 25%-75% of the target nail altered as a result of onychomycosis
* Signed written informed consent

Exclusion criteria

* Proximal subungual onychomycosis
* Patient who has been previously randomized to treatment in the phase III study K70-2 investigating K101
* Other conditions known to cause abnormal nail appearance
* Use of topical (1 month before screening) and/or systemic (3 months before screening) antifungal medication.
* Participation in another clinical study with an investigational drug or device during the previous 4 weeks before enrolment.
* Known allergy to any of the tested treatment products

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing at least some improvement of the target nail (scoring 2 or more according to Global Assessment Scale) after 8 weeks treatment.